CLINICAL TRIAL: NCT05335148
Title: Evaluate the Safety of Colchicine for Treatment and Prevention of Radiation-Induced Dermatitis
Brief Title: Study to Evaluate the Safety of Colchicine
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Bruce G Haffty, Associate Vice Chancellor Cancer Programs Professor and Chairman Department of Radiation Oncology, Rutgers, The State University of New Jersey
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 032112; Pro2022000357 (Other: Rutgers, The State University of New Jersey)
Record Dates: First submitted 2022-04-13; First posted 2022-04-19 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Radiation Therapy
Keywords: Radiation therapy; Dermatitis; Low-dose colchicine
MeSH Terms: conditions — Dermatitis | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: Perform a phase I study for evaluating the safety of oral colchicine in preventing and treating radiation-induced dermatitis among head and neck cancer patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care arm - placebo colchicine pill (No Intervention): The standard of care arm will receive a placebo colchicine pill once a day
- Experimental arm - oral colchicine once a day (Experimental): The experimental arm will receive 0.6 mg of oral colchicine once a day
  Interventions: Drug: oral colchicine(0.6 mg) once a day

INTERVENTIONS:
Drug: oral colchicine(0.6 mg) once a day — The standard of care arm will receive a placebo colchicine pill once a day
  Arms: Experimental arm - oral colchicine once a day

SUMMARY:
Currently, there are no approved medications for the prevention and treatment of radiation-induced dermatitis, or skin discoloration/burning due to radiation therapy, because there is little evidence to guide treatment.

The purpose of the research is to better understand the factors associated with radiation-induced dermatitis and to explore the efficacy of low-dose colchicine in reducing the proportion of patients with radiation-induced dermatitis who undergo radiation treatment for head and neck cancer. If you take part in the research, you will be asked to take 0.6 mg once a day by mouth. The participants time in the study will take less than a minute a day to take the pill and 20 minutes to complete survey questions during follow-up visits.

DETAILED DESCRIPTION:
A phase I study for evaluating the safety of oral colchicine in preventing and treating radiation-induced dermatitis among head and neck cancer patients who will receive RT for HNC. Prior to receiving RT, each subject will be receiving either the standard of care or low-dose oral colchicine (No randomization). There will be a comparison of the proportion of radiation-induced dermatitis in the two study arms. The individuals in the standard of care arm will receive a placebo colchicine pill once a day. Those who are in the experimental arm will receive 0.6 mg of oral colchicine once a day. The primary endpoint is the safety and tolerability of oral colchicine. The proportions of grade 2-4 radiation-induced dermatitis at the end of Radiation therapy (RT) and at the first follow-up three-four weeks post-treatment in these two study arms are the secondary study endpoints. In addition, pain, erythema, and health-related quality-of-life will be evaluated.

The study subjects will receive radiation therapy (RT) as scheduled and will meet with their clinicians for their follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Eight years or older with HNC diagnosis confirmed histologically

  o Stage 1-3 HNC pathologically confirmed diagnosis of squamous cell carcinoma of the oropharynx, larynx, hypopharynx, nasopharyngeal, or oral cavity
* Plan to receive radiotherapy (>60 Gy), chemo-irradiation or bio-radiation either as primary or as a post-operative treatment to the head and neck region
* Eastern Cooperative Oncology Group Performance Status (ECOGPS) performance status 0 or 1
* Comply with the study protocol
* Capable of signing a written informed consent

Exclusion Criteria:

* An allergy, intolerance, or contraindication to colchicine
* Current treatment with colchicine for medical conditions, e.g. gout and Familial Mediterranean Fever (FMF)
* Estimated glomerular filtration rate (GFR) < 55 ml/min since colchicine should not be given
* Severe liver disease or current aminotransferase levels of more than 1.5 times the upper limit of the normal range
* Previous irradiation to the head and/or neck region
* Distant metastatic disease or locally recurrent disease
* Pre-existing skin rashes, ulcerations, or open wounds in the treatment area
* Known allergic and other systemic skin diseases even when not directly affecting irradiated fields
* Substance abuse, medical conditions, and/or social issues that would limit conduct or follow-up in the research study, in the opinion of the investigator
* Any condition that is unstable or could affect the safety of the patient and their compliance in the study as judged by the investigator
* Using high doses of non-steroidal anti-inflammatory drugs
* Pregnant and lactating women
* Psychiatric illness that would prevent the patient from giving informed consent
* Taking cetuximab or other radiosensitizing agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain - Visual Analogue Scale (VAS) | 10 weeks
  Pain (within radiation fields): assessed before radiotherapy, weekly during radiotherapy, and at the end of treatment with the visual analogue scale (VAS) (from 0 = no pain to 100 = maximum pain)

SECONDARY OUTCOMES:
Erythema - Common Toxicity Criteria for Adverse Events (CTCAE) | 10 weeks
  The National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) scale defines acute skin reactions to radiation occurring within the 90 days after therapy.
  Grade 1: faint erythema or dry desquamation. Arising within the first two to four weeks of treatment, these reactions cause skin redness, warmth, and a rash-like appearance. The patient may complain that their skin feels tight or sensitive.
  Grade 2: moderate to brisk erythema; patchy, moist desquamation usually confined to skin folds or creases. Moderate edema, dryness, pruritus, and flaking of skin layers (dry desquamation) also may occur.
  Grade 3: moist desquamation in areas other than creases and skinfolds. Bleeding may arise from minor trauma, such as abrasion.
  Grade 4: life-threatening consequences, such as full-thickness skin ulcers, necrosis, and spontaneous bleeding.
  Grade 5: death.

OTHER OUTCOMES:
Health-Related Quality-of-Life - Questionnaire | 10 weeks
  Health-related quality of life (HRQOL) measured before, during, and after Radiation therapy, with a validated HRQOL questionnaire, European Organization for Research and Treatment of Cancer (EORTC)
Health-Related Quality-of-Life - Quality of Life Questionnaire | 10 weeks
  Treatment of Cancer European Organization for Research and Treatment of Cancer (EORTC). A validated questionnaire developed to assess the quality of life of cancer patients.
  Quality of Life Questionnaire Core Module (QLQ-C30) version- 3.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Haffty, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (3):
- United States (3):
  - RWJBarnabas Health - Cooperman Barnabas, Livingston, New Jersey
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers, The State University of New Jersey Board Contact:, New Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: No